CLINICAL TRIAL: NCT06323551
Title: The Effect of Mother's Smell and Breast Milk Smell on Pain and Crying Time During Heel Blood Collection in Newborns
Brief Title: The Effect of Mother's Smell and Breast Milk Smell on Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Atiye Karakul, Assoc. prof., Tarsus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023/50
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Newborn; Vitality; Pain; Crying
Keywords: Crying Time; pain; newborn
MeSH Terms: conditions — Pain; Crying

STUDY DESIGN:
Intervention Model Description: randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mother's Smell (Experimental): In the study group that will be made to smell the mother's scent; The mother of each baby whose heel blood will be taken will be given a specially made cover made of 100% cotton yarn, sterilized the day before, and the mother will be asked to put the cover on her bare skin (on her bare skin) after the shower and to keep the cover on the mother's chest for one night (8 hours). one). It will be placed 15 cm away from the baby and smelled 5 minutes before and 5 minutes after the heel prick attempt (1,4). The baby's pain score will be evaluated by the observing nurse according to the NIPS pain scale 5 minutes before, during and 5 minutes after the procedure.
  Interventions: Other: Mother's Smell
- Mother's Breast Milk Smell (Experimental): In the study group that will be made to smell the scent of breast milk, the procedures for the scent of the mother will be carried out in the same way, and 20 drops of each baby's own mother's milk will be dropped onto the diaper (4). The cover, which has the scent of breast milk, will be placed 15 cm away from the baby and allowed to smell it from 5 minutes before to 5 minutes after the heel prick blood collection attempt. The baby's pain score will be evaluated by the observing nurse according to the NIPS pain scale 5 minutes before, during and 5 minutes after the procedure.
  Interventions: Other: Mother's Breast Milk Smell
- Control (No Intervention): Routine care will be provided to the control group and no intervention will be applied.

INTERVENTIONS:
Other: Mother's Smell — The mother of each baby whose heel blood will be taken will be given a specially made cover made of 100% cotton yarn, sterilized the day before, and the mother will be asked to put the cover on her bare skin (on her bare skin) after the shower and to keep the cover on the mother's chest for one night (8 hours). one).
  Arms: Mother's Smell
Other: Mother's Breast Milk Smell — In the study group that will be made to smell the scent of breast milk, the procedures for the scent of the mother will be carried out in the same way, and 20 drops of each baby's own mother's milk will be dropped onto the diaper.
  Arms: Mother's Breast Milk Smell

SUMMARY:
The research was planned as a randomized controlled study to investigate the effect of breast milk smell and mother's smell applied while heel blood was taken to term babies in the Mersin City EAH Neonatal Intensive Care Unit between October and December 2023, on acute pain and crying duration. During the heel prick procedure, which is routinely performed in the neonatal intensive care unit, no pharmacological/non-pharmacological method will be applied to the control group to reduce the baby's pain before, during and after the heel prick. The baby's pain score will be evaluated by the observing nurse according to the NIPS pain scale 5 minutes before, during and 5 minutes after the procedure.

In the study group that will be made to smell the mother's scent; The mother of each baby whose heel blood will be taken will be given a specially made cover made of 100% cotton yarn, sterilized the day before, and the mother will be asked to put the cover on her bare skin (on her bare skin) after the shower and to keep the cover on the mother's chest for one night (8 hours). It will be placed 15 cm away from the baby and smelled 5 minutes before and 5 minutes after the heel prick attempt. The baby's pain score will be evaluated by the observing nurse according to the NIPS pain scale 5 minutes before, during and 5 minutes after the procedure.

DETAILED DESCRIPTION:
The research was planned as a randomized controlled study to investigate the effect of breast milk smell and mother's smell applied while heel blood was taken to term babies in the Mersin City EAH Neonatal Intensive Care Unit between October and December 2023, on acute pain and crying duration.

The population of the research will consist of all-term babies followed in the Mersin Şehir EAH neonatal intensive care unit.

As a result of Power analysis (G*Power 3.1.9.2) based on Akcan and Polat's (2015) study titled "The effect of breast milk, amniotic fluid and lavender scent on pain during invasive procedures in newborns"; In the evaluation made according to the NIPS score, when the Effect Size was taken as 0.619, the minimum number of samples for each group determined for Power: 0.95 was determined as 28 newborns. Considering the case losses, it was planned to include 30 newborns in each group.

Randomization: In the study, 60 newborns in the sample will be randomly assigned to the control and breast milk scent groups. Random assignments will be made using a computer program to determine the group in which the newborns will be placed (https://www.randomlists.com/team-generator).

During the heel prick procedure, which is routinely performed in the neonatal intensive care unit, no pharmacological/non-pharmacological method will be applied to the control group to reduce the baby's pain before, during, and after the heel prick. The baby's pain score will be evaluated by the observing nurse according to the NIPS pain scale 5 minutes before, during and 5 minutes after the procedure.

In the study group that will be made to smell the mother's scent; The mother of each baby whose heel blood will be taken will be given a specially made cover made of 100% cotton yarn, sterilized the day before, and the mother will be asked to put the cover on her bare skin (on her bare skin) after the shower and to keep the cover on the mother's chest for one night (8 hours). It will be placed 15 cm away from the baby and smelled 5 minutes before and 5 minutes after the heel prick attempt. The baby's pain score will be evaluated by the observing nurse according to the NIPS pain scale 5 minutes before, during and 5 minutes after the procedure.

In the study group that will be made to smell the scent of breast milk, the procedures for the scent of the mother will be carried out in the same way, and 20 drops of each baby's own mother's milk will be dropped onto the diaper. The cover, which has the scent of breast milk, will be placed 15 cm away from the baby and allowed to smell it from 5 minutes before to 5 minutes after the heel prick blood collection attempt. The baby's pain score will be evaluated by the observing nurse according to the NIPS pain scale 5 minutes before, during and 5 minutes after the procedure.

During the study, all factors that may affect the pain level of babies in the intervention and control groups will be standardized. In this context, attention will be paid to factors such as ensuring that the procedure is performed when the baby is not crying, applying a 2-minute waiting period if the baby is crying, and ensuring that the heel blood is taken by experienced and always the same nurse.

ELIGIBILITY:
Inclusion Criteria:

* Term newborns receiving treatment in Mersin City Training and Research Hospital Neonatal Intensive Care Service,
* Postnatal 1-15. Newborns on their day,
* Newborns who have not previously used any pharmacological or non-pharmacological method for pain management,
* Newborns with an Apgar score of 8 points or more at the 1st and 5th minutes,
* Not having undergone a surgical procedure,
* Does not have any health problems,
* Patients whose families approve the informed consent form.

Exclusion Criteria:

* Born before 37 weeks of gestation, receiving treatment in the Neonatal Intensive Care Service at Mersin City Training and Research Hospital,
* Sedation area
* Except for major congenital anomaly
* Older than the 15th postnatal day,
* Having a major anomaly or disease detected antenatally,
* Patients with comorbid diseases such as perinatal asphyxia, bronchopulmonary dysplasia, intraventricular hemorrhage, necrotizing enterocolitis, congenital heart disease and similar diseases,
* Patients whose families do not give consent will not be included in the study.

Ages: 1 Day to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale | 1 day
  The Neonatal Infant Pain Scale was developed at Children's Hospital of Eastern Ontario. The Scale assesses six behavioral indicators in response to painful procedures in preterm newborns.The total score varies between 0 and 7 points, and a higher score indicates more pain

SECONDARY OUTCOMES:
criying time | 1 day
  During the procedure, crying time will be measured with a stopwatch.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus State Hospital, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kucuk Alemdar D, Kardas Ozdemir F. Effects of Having Preterm Infants Smell Amniotic Fluid, Mother's Milk, and Mother's Odor During Heel Stick Procedure on Pain, Physiological Parameters, and Crying Duration. Breastfeed Med. 2017 Jun;12:297-304. doi: 10.1089/bfm.2017.0006. Epub 2017 Apr 17. PMID 28414516
- [Background] Gellrich J, Breuer AS, Han P, Guducu C, Hummel T, Schriever VA. Central Nervous System Processing of Floral Odor and Mother's Milk Odor in Infants. Chem Senses. 2021 Jan 1;46:bjab024. doi: 10.1093/chemse/bjab024. PMID 34003211
- [Background] 3. Yigit, S., Ecevit, A., & Koroglu, O. A. (2018). Guidelines for pain and treatment in the newborn period. Turkish Neonatology Association, 53, 161-171.
- [Background] Cakirli M, Acikgoz A. A Randomized Controlled Trial: The Effect of Own Mother's Breast Milk Odor and Another Mother's Breast Milk Odor on Pain Level of Newborn Infants. Breastfeed Med. 2021 Jan;16(1):75-81. doi: 10.1089/bfm.2020.0222. Epub 2020 Oct 20. PMID 33085532
- [Background] 5. Çöçelli, L. P., Bacaksız, B. D., & Ovayolu, N. (2008). The nurse factor in pain therapy. European Journal of Therapeutics, 14(2), 53-58.
- [Background] Lan HY, Yang L, Lin CH, Hsieh KH, Chang YC, Yin T. Breastmilk as a Multisensory Intervention for Relieving Pain during Newborn Screening Procedures: A Randomized Control Trial. Int J Environ Res Public Health. 2021 Dec 10;18(24):13023. doi: 10.3390/ijerph182413023. PMID 34948633
- [Background] Beker F, Opie G, Noble E, Jiang Y, Bloomfield FH. Smell and Taste to Improve Nutrition in Very Preterm Infants: A Randomized Controlled Pilot Trial. Neonatology. 2017;111(3):260-266. doi: 10.1159/000450883. Epub 2016 Dec 1. PMID 27902988
- [Background] Baudesson de Chanville A, Brevaut-Malaty V, Garbi A, Tosello B, Baumstarck K, Gire C. Analgesic Effect of Maternal Human Milk Odor on Premature Neonates: A Randomized Controlled Trial. J Hum Lact. 2017 May;33(2):300-308. doi: 10.1177/0890334417693225. Epub 2017 Mar 27. PMID 28346843
- [Background] 9. Akcan E. Yenidoğanlarda Topuk Kanı Alma Sırasında Oluşan Ağrıya Amniyotik Sıvı, Anne Sütü Ve Lavanta Kokusunun Etkisi (tez). Kayseri: Erciyes Üniversitesi; 2014.